CLINICAL TRIAL: NCT06731699
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of FD-001 in Patients with Relapsed or Refractory Hematological Malignancies.
Brief Title: A Phase 1 Study of FD-001 in Recurrent /Refractory (R/R)AML/NHL/MM/MDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu FenDi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-MD-23001
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: AML; NHL
Keywords: FD-001; AML; NHL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FD-001 (Experimental)
  Interventions: Drug: FD-001

INTERVENTIONS:
Drug: FD-001 — The initial dose was 0.4mg, and subsequent doses of 0.8mg, 1.6mg, 2.4mg, 3.2mg, and 4.0mg were proposed to be administered in a progressive manner using the "rapid titration" method combined with the traditional "3+3" experimental design. The trial process consists of three periods: screening period, treatment period, and follow-up period. The screening period lasted from D-28 to D-1 for treatment (DLT observation period): during this time frame, there was a single administration period (C0D1-C0D4) where oral administration occurred on day one followed by safety observations on days two to four; as well as multiple administration period one (C1D1-C1D28) where oral administration took place on days one to two and seven to nine with rest periods in between. The drug is available in capsule form.

SUMMARY:
This is a single-arm, open-label, dose-escalation and dose-expansion phase I clinical trial aimed at assessing the safety, tolerability, pharmacokinetic/pharmacodynamic profile, and preliminary efficacy of FD-001 capsules in the treatment of recurrent/refractory hematologic malignancies(AML/MDS/NHL/MM). The trial consists of two phases: the initial phase (dose escalation) and the subsequent phase (dose expansion). The primary objectives are to evaluate the safety and tolerability of FD-001 in subjects with recurrent/refractory hematologic tumors and determine the maximum tolerated dose (MTD) as well as the recommended Phase II dose (RP2D) for FD-001 in this patient population.

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose-escalation and dose-expansion phase I clinical trial aimed at assessing the safety, tolerability, pharmacokinetic/pharmacodynamic profile, and preliminary efficacy of FD-001 capsules in the treatment of recurrent/refractory hematologic malignancies(AML/MDS/NHL/MM).The trial process consists of three periods: the screening period, the treatment period, and the follow-up period. The screening period occurred from D-28 to D-1. The treatment period (DLT observation period) includes a single administration phase (C0D1-C0D4) (oral administration on D1, followed by safety observation from D2-D4), as well as multiple administration phase 1 (C1D1-C1D28) (oral administration on D1-D2 and D7-D9, with withdrawal for the remaining time). Blood samples were collected in the first cycle (C1D1~C1D28) for PK study, and part of the PK test blood samples may be used for metabolite identification.After completion of the DLT evaluation, subjects without intolerable toxicity may enter the maintenance treatment period if determined by the investigator that continued treatment outweighs risks. The maintenance treatment period lasts for 28 days per cycle (CND1-CND28), with oral administration on D1-D3 and D8-D10 per cycle, while withdrawing for the rest of the time.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to voluntarily participate in this clinical study; possess a comprehensive understanding of, provide consent for, and sign the written informed consent form (ICF) for this study; demonstrate willingness to adhere to and complete all study procedures.
2. Age range from 18 to 80 years (inclusive), with no gender restrictions.
3. ECOG performance status ≤2 (refer to Appendix 1).
4. Expected minimum survival period of at least 3 months.
5. Patients diagnosed with hematological malignancies confirmed through pathological and/or cytological examinations, who have either failed or not received standard treatment due to lack of efficacy or intolerance. This includes patients with recurrent/refractory conditions.
6. Presence of at least one measurable lesion:

   * For AML: bone marrow containing more than 5% primitive/immature cells (excluding regeneration after consolidation chemotherapy).
   * For MDS: bone marrow aspirate or biopsy pathological examination revealing less than 20% primitive cells.
   * For MM: meeting any of the following criteria:

     1. Monoclonal protein detected in blood ≥1 g/dL (10g/L) through serum protein electrophoresis.
     2. Urine monoclonal protein ≥200 mg over a span of 24 hours.
     3. If monoclonal protein is undetectable in blood or urine, affected-to-unaffected serum FLC ratio should be ≥100 (with affected serum FLC level being ≥100 mg/L).
   * For NHL: presence of measurable lesions identified by CT, PET-CT, or PET-MRI scans such as lymph node lesions with major axis >1.5 cm or extranodal lesions with major axis >1.0 cm); CLL/SLL: peripheral blood monoclonal lymphocytes ≥5.0×10^9/L; WM: IgM >2×ULN.
7. Adverse effects resulting from previous anti-cancer therapy should have recovered to grade ≤1 (continuous hair loss excluded along with laboratory tests specified in criterion 8).
8. With sufficient organ function support, all the following criteria must be met during the laboratory tests in the screening period:

   * The white blood cell (WBC) count should be less than or equal to 30×10^9/L before the first use of the investigational drug; (This criterion is only applicable to AML and MDS, and the use of hydroxyurea to lower the white blood cell count is permitted.) The absolute neutrophil count (ANC) should be greater than or equal to 1.0×10^9/L before the first use of the investigational drug, and it can be relaxed to 0.75×10^9/L in the case of bone marrow infiltration; the platelet count (PLT) should be greater than or equal to 70×10^9/L before the first use of the investigational drug, and it can be relaxed to 50×10^9/L in the case of bone marrow infiltration; the hemoglobin (HB) level should be greater than or equal to 70 g/L before the first use of the investigational drug, and it can be relaxed to 60 g/L in the case of bone marrow infiltration (This criterion is only applicable to MM and NHL; It is required that this test was not conducted within 7 days before blood collection after the administration of G-CSF (or GM-CSF), erythropoietin, thrombopoietin treatment or component blood transfusion)

Exclusion Criteria:

1. Within 4 weeks prior to the first dose of the study drug or within 5 half-lives (whichever is shorter), the subject has received anti-cancer therapy, including chemotherapy, immunotherapy, targeted therapy (excluding hydroxyurea therapy and prophylactic intrathecal injection of chemotherapy drugs); received radiation therapy within 2 weeks; received anti-cancer therapy with Chinese herbal medicine within 2 weeks;
2. Chronic myeloid leukemia (CML) with BCR/ABL positivity;
3. The subject has central nervous system malignant tumor infiltration;
4. The subject has another malignant tumor at the same time (excluding IB stage or lower-stage cervical cancer that has been cured, non-invasive basal cell or squamous cell skin cancer, and other malignant tumors that have achieved complete remission (CR) >10 years and >5 years, respectively);
5. Within 4 weeks prior to the first dose of the study drug, the subject has received an active or attenuated live vaccine;
6. The subject has a history of clear alcohol and drug abuse; a history of severe allergies in the past, or is allergic to any component of the study drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Phase Ⅰa:Dose limiting toxicity(DLT) | From enrollment to the end of treatment at 32 days
  DLT are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly,probably or definitely related to study drug administration
Phase Ⅰa:Maximum tolerated dose(MTD) | From enrollment to the end of treatment at 32 days
  MTD is defined as the highest dose level at which no more than 1 in 3 participants experienced a DLT during the first cycle
Phase Ⅰb:Recommended Phase Ⅱ Dose(RP2D) | From enrollment to the end of treatment at 32 days
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase Ⅱ study,based on safety,tolerability,efficacy,PK,and PD data collected during the dose escalation study of FD-001.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  ORR is defined as the percentage of participants,who has a CR or PR
Cmax | Hour 0,0.5,1,2,3,4,6,12,24,48,72hours post-dose on single dose;Hour 0 of day 7,day8 on multiple dose and hour 0,0.5,1,2,3,4,6,12,24,48,72hours post-dose on multiple dose of day 9
  Maximum serum concentration(Cmax) of FD-001 will be investigated
Tmax | Hour 0,0.5,1,2,3,4,6,12,24,48,72hours post-dose on single dose;Hour 0 of day 7,day8 on multiple dose and hour 0,0.5,1,2,3,4,6,12,24,48,72hours post-dose on multiple dose of day 9
  To characterize the pharmacokineties of FD-001by assessment of time to reach maximum plasma concentration
Area Under the Curve (AUC)0-t | Hour 0,0.5,1,2,3,4,6,12,24,48,72hours post-dose on single dose;Hour 0 of day 7,day8 on multiple dose and hour 0,0.5,1,2,3,4,6,12,24,48,72hours post-dose on multiple dose of day 9
  To characterize the pharmacokinetics of FD-001 by assessment of area under the plasma concentration time curve from zero to infinity
T1/2 | Hour 0,0.5,1,2,3,4,6,12,24,48,72hours post-dose on single dose;Hour 0 of day 7,day8 on multiple dose and hour 0,0.5,1,2,3,4,6,12,24,48,72hours post-dose on multiple dose of day 9
  To characterize the pharmacokinetics of FD-001 by assessment of the duration required for the peak plasma concentration to be reduced by half

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China